CLINICAL TRIAL: NCT02964364
Title: China Takayasu Arteritis Registry (CTA Registry)
Status: Recruiting | Type: Observational
Sponsor: Aimin Dang (Other)
Responsible Party: Sponsor-Investigator, Aimin Dang, Fuwai Hospital, Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Other Study IDs: NSFC 30770859
Record Dates: First submitted 2016-08-21; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-09

CONDITIONS: TAKAYASU ARTERITIS
Keywords: TAKAYASU ARTERITIS
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Takayasu arteritis (TA) is a chronic large-vessel vasculitis that mainly affects the aorta and its major branches. The epidemiology and pathophysiology of TA is still unclear in China, although many studies have been done. Our previous study supporting by National Natural Science Foundation of China indicated the cytokines such as hs-CRP, NT-proBNP and tumor necrosis factor-alpha (TNF-α) can be used to monitor TA activity, and HLA gene alleles were associated with TA in Chinese han population. Further investigations with larger samples are needed to fully understand the a pathophysiology of TA. The purpose of this study is to build a Chinese national registry system for TA to obtain real-world information, such as current status of characteristics, diagnosis, disease activity, the severity of disease, treatment and outcomes of Chinese TA patients. To analysis and development of effective disease monitoring and treatment strategies.

DETAILED DESCRIPTION:
Takayasu arteritis (TA) is a chronic vasculitis that causes inflammation of the aorta and its main branches and is characterized by adventitial thickening and cellular infiltration of the tunica media, with local destruction of vascular smooth muscle cells and elastin. The disease is very rare but most commonly occurs in China. In the last decade, the results of our study indicated that HLA-DPB1, HLA-DQA1, HLA-DQB1 and HLA-DRB1 gene alleles were associated with TA in Chinese Han population. And the clinical features of patients with TA were analyzed. The cytokines such as hs-CRP, NT-proBNP and tumor necrosis factor-alpha (TNF-α) can be used to monitor TA activity. But there are still many unknown fields in TA, such as the epidemiology and pathophysiology. This study is to build a Chinese national registry system for TA to obtain real-world information, such as current status of characteristics, diagnosis, disease activity, the severity of disease, treatment and outcomes of Chinese TA patients. To analysis and development of effective treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age at disease onset < 40 years. (Development of symptoms or findings related to Takayasu arteritis at age <40 years)
* Claudication of extremities. (Development and worsening of fatigue and discomfort in muscles of 1 or more extremity while in use, especially the upper extremities)
* Decreased brachial artery pulse. (Decreased pulsation of 1 or both brachial arteries)
* BP difference >10 mm Hg. (Difference of >10 mm Hg in systolic blood pressure between arms)
* Bruit audible on auscultation over 1 or both subclavian arteries or abdominal aorta.
* Arteriogram abnormality. (Arteriographic narrowing or occlusion of the entire aorta, its primary branches, or large arteries in the proximal upper or lower extremities, not due to arteriosclerosis, fibromuscular dysplasia, or similar causes; changes usually focal or segmental)

Exclusion Criteria:

* Vessel lesions that could be entirely due to atherosclerosis.
* Giant cell arteritis or other infectious forms of large vessel vasculitis.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with TA. Participants will have disease in various stages and of different duration.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mortality of the patients with TA | 10 years （2016-2026）
  All-caused death at 10 years.

SECONDARY OUTCOMES:
The rate of the major cardiac and cerebrovascular events | 10 years （2016-2026）
  the major cardiac and cerebrovascular events (MACCE) defined as the composite of all heart failure, all stroke, all myocardial infarction (MI), or any revascularization at 10 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Medical clinical data base